CLINICAL TRIAL: NCT00399854
Title: Clinical Study for Evaluation of the Efficacy of Mechanical Massage by Endermologie (Dhermia® - Industra Mecânica Fina Ltda) in Treatment of Cellulite and Body Contouring
Brief Title: Evaluation of the Efficacy of Endermologie in Treatment of Cellulite and Body Contouring
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hexsel Dermatology Clinic (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02CBED0501
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2006-11-15 (Estimated); Status verified 2006-11

CONDITIONS: Cellulite; Body Contouring
MeSH Terms: conditions — Cellulite

INTERVENTIONS:
Device: Dhermia® - Industra Mecânica Fina Ltda

SUMMARY:
The purpose of this study is to perform a clinical assessment of the efficacy of the device DHERMIA® (Industra Mecânica Fina Ltda)in the treatment of cellulite and body contouring

DETAILED DESCRIPTION:
The present study is a clinical, opened trial and single-center.

The patients were treated by endermologie device. Mechanical massage were performed for 12 weeks in a total of 24 treatment sessions: twice a week.

A set of photographs were took at visit 1 (baseline), visit 2, 3 and 4 with standardized positions and lighting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent;
2. Subjects agreeing to take part of all procedures of the study (including mechanical massage, photographs), after being fully informed on the objectives and nature of the investigations;
3. Female subjects between 25-45 years;
4. Subjects presenting with cellulite grades I-III on buttocks and thighs;
5. Medical history and physical examination which, based on the investigator's opinion, do not prevent the patient from taking part in the study and use the device under investigation;
6. Female subjects of childbearing age should present a negative urine pregnancy test and should be using an effective contraceptive method (3 months before the enrollement untill the end of the study);
7. Body Mass Index (BMI = weight/height2) beetwen 20,0-25,0 and 25,0-29,9;
8. Availability of the subject throughout the duration of the study (90 days);
9. Availability of the subject in maintaining a stable weight during the study (variation less than 2 kg)
10. Subjects with sufficient schooling and awareness to enable them to cooperate to the degree required by this protocol.

Exclusion Criteria:

1. Pregnant women or women intending to become pregnant during the study (next 3 months);
2. BMI superior 30,0;
3. Subjects with diabetes mellitus, cardiac insufficiency, asthma, or bronchitis;
4. Subjects participating in other clinical trials;
5. Subjects with neoplastic disorders, uncontrolled thyroid disorders or uncontrolled hypertension;
6. Subjects with coagulation disorders, using anticoagulants or tendency of bruises;
7. Subjects with vascular disorders (phlebitis or varicose veins) in the area to be treated;
8. Any prior aesthetic surgery affecting the area to be treated (liposuction, Subcision®), 3 months before the study, that may interfere with results;
9. Any other prior anti-cellulite treatment or body measures treatment, 30 days prior to the study;
10. Subjects with inflammation or active infection in the area to be treated.
11. Subjects with a history of adverse effects, which in the investigator's opinion should prevent the patient from participating in the study;
12. Patients with cutaneous or vascular alterations, that difficult visualization and documentation of cellulite;
13. Subjects with a history of medical treatment non-adherence or showing unwillingness to adhere to the study protocol;
14. Subjects who can not come to the visits (one missing visit/ month is allowed);
15. Subjects intending to initiate any intensive sport;
16. Subjects using analgesics, non-hormonal antiinflammatories, antihistaminics, corticosteroids, or diuretics;
17. Subjects tanned, or intending to expose the area of study to sun, artificial UV, or self-tanning during the study;
18. Any condition that, in the opinion of the investigator, can compromise the evaluation of the study.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45
Dates: Start 2006-03; Study Completion 2006-07

PRIMARY OUTCOMES:
Assessment of effectiveness of treatment based on current classification of cellulite and evaluation of the corporal measures

SECONDARY OUTCOMES:
Assessment of subject's satisfaction
Visual assessments of the treated area before and after treatment
Safety analysis

CONTACTS AND LOCATIONS:
Overall Officials: Doris Hexsel, MD, Study Director — Hexsel Dermatology Clinic